CLINICAL TRIAL: NCT00642135
Title: Efficacy and Tolerance of Ophthalmic Insert Mydriasert® Versus Reference Treatment (Phenylephrine and Tropicamide Eyedrops) in Premature Newborns, Neonates and Infants Justifying a Mydriasis for a Bilateral Diagnosis Fundus
Brief Title: CLAIR -FO: Clinical Trial of Ophthalmic Insert Mydriasert® Versus Reference Treatment
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The total number of patients has been reached.
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ioltech (Industry)
Responsible Party: Mathieu QUINTIN, Department Clinical Research of Developpement
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P050308; réf Afssaps : 437-050883-LB/GG; Eudract : 2005-004418-33
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2006-01

CONDITIONS: Retinal Anomalies; Premature Birth
Keywords: premature; neonates; infants; children; Mydriasert®; mydriasis; fundus; Tropicamide; Phenylephrine; clinical trial; Infant; premature newborns; bilateral diagnosis fundus
MeSH Terms: conditions — Premature Birth; Mydriasis | interventions — Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Premature newborns and neonates treated using Phenylephrine and tropicamide eyedrops
  Interventions: Drug: phenylephrine and tropicamide eyedrops
- 2 (Active Comparator): Premature newborns and neonates treated using insert Mydriasert®
  Interventions: Drug: Mydriasert®

INTERVENTIONS:
Drug: Mydriasert® — Premature newborns and neonates treated using ophthalmologic insert Mydriasert®
  Arms: 2
Drug: phenylephrine and tropicamide eyedrops — Premature newborns and neonates treated using reference treatment (association of Phenylephrine and tropicamide eyedrops)
  Arms: 1

SUMMARY:
Pupillary dilation to perform a fundus in premature newborns and neonates is often difficult to obtain, because of the non mature iris sphincter. The fundus is essential to detect retinal anomalies (as retinopathy of prematurity or chorioretinal or disk anomalies). The aim of the study is to obtain a satisfactory degree of mydriasis with a minimal dose of two mydriatic treatments, with an optimal duration and a good tolerance of the drugs. The study will evaluate the mydriasis in premature newborns, neonates and infants justifying a mydriasis for a bilateral diagnosis fundus, using ophthalmic insert Mydriasert® versus reference treatment (association of phenylephrine and tropicamide eyedrops). Ophthalmic insert Mydriasert® can control drug dispensation and decrease the number of nurse interventions to obtain mydriasis in patients.

DETAILED DESCRIPTION:
The aim of the study is to obtain a satisfactory degree of mydriasis with a minimal dose of two mydriatic treatments, with an optimal duration and a good tolerance of the drugs. The study will evaluate the mydriasis in premature newborns, neonates and infants justifying a mydriasis for a bilateral diagnosis fundus, using ophthalmic insert Mydriasert® versus reference treatment (association of phenylephrine and tropicamide eyedrops). Ophthalmic insert Mydriasert® can control drug dispensation and decrease the number of nurse interventions to obtain mydriasis in patients.

ELIGIBILITY:
Inclusion Criteria:

* Premature newborns, neonates and infants of less 18 months-old indoor in the neonatology clinical department of Robert Debre Hospital with cardiologic monitoring
* Presenting a risk of retinopathy of prematurity or fundus anomaly (chorioretinal and/or disk anomalies).
* Needing a bilateral fundus
* Parents, tutor or legal representing of the patient had been informed of objectives of the study and had given their written consent.
* Covered by French social security or CMU

Exclusion Criteria:

* Neonates of less 1000g at inclusion
* Premature newborn of less 30 weeks of gestational age at inclusion
* Contra-indication to one of the evaluated drugs
* Any treatment that could provoke a dangerous drug interaction for the patient if associated with one of the drug of the study
* Anatomical predisposition to glaucoma, hypertension or any other contra-indication noted by the physician

Max Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2006-01; Primary Completion 2008-02 (Estimated); Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Mydriasis larger than 5,5 mm with absence of photometer reflex to get a satisfactory fundus. | 75 minutes

SECONDARY OUTCOMES:
Frequency of the nurse intervention to obtain the mydriasis | during 215 minutes maximum
Calculation of the dose of active drugs administrated | one day
Local and systemic clinical tolerance | one day
Occurrence of adverse reactions | one day
Stability of a mydriasis of good quality at T+195 | at T+195 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Dominique BREMOND GIGNAC, MD, Principal Investigator — Hôpital Robert Debré, APHP, France
Locations (1):
- Hôpital Robert Debré, Paris, France